CLINICAL TRIAL: NCT04426370
Title: The Effects of Social Role Participation on Life Quality in Rheumatoid Arthritis Patients
Brief Title: The Effects of Social Role Participation on Life Quality
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gul Devrimsel, Assoc. Prof., Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: gd230863
Record Dates: First submitted 2020-06-07; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Social Interaction
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: 100 rheumatoid arthritis patients (age from 20 to 70 years)
  Interventions: Other: Observational
- Control: 95 healthy volunteer
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Physical examination and questionnaires

SUMMARY:
The study was carried out among 100 RA patients (age from 20 to 70 years) by fulfilling the American College of Rheumatology 1987 revised criteria admitted to our outpatient clinic. RA patients were compared with 95 healthy volunteer control group. Participants were asked to complete interview based questionnaires regarding pain, life quality, and social role participation to obtain additional information during the interview to participate in the study in 20 min.

DETAILED DESCRIPTION:
The study was carried out among 100 RA patients (age from 20 to 70 years) by fulfilling the American College of Rheumatology 1987 revised criteria admitted to our outpatient clinic. RA patients were compared with 95 healthy volunteer control group. Healthy volunteers were recruited from the partners next to the patients who came to our outpatient clinic for examination. The same physician carried out the physical examinations on all participations and conducted a interview, acquiring information on age, gender, body mass index (BMI), marriage status, living alone, working, and education. Participants were asked to complete interview based questionnaires regarding pain, life quality, and social role participation to obtain additional information during the interview to participate in the study in 20 min. Examinations took place at the our outpatient clinic. This study did not include all participants who had accompanying of other rheumatic diseases, musculoskeletal diseases, the presence of another chronic disease, cancer.

ELIGIBILITY:
Inclusion Criteria:The study was carried out among RA patients (age from 20 to 70 years) by fulfilling the American College of Rheumatology 1987 revised criteria admitted to our outpatient clinic -

Exclusion Criteria:This study did not include all participants who had accompanying of other rheumatic diseases, musculoskeletal diseases, the presence of another chronic disease, cancer.

-

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 100 RA patients and 95 healthy volunteer control
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Social role participation | 4 months
  Social role participation questionnaire